CLINICAL TRIAL: NCT05220644
Title: Management of Pain Respiratory Distress at the End of Life in Newborn Palliative Care in the
Brief Title: Management of Pain Respiratory Distress at the End of Life in Newborn Palliative Care in the Delivery Room
Acronym: PALLI-ACC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8339
Record Dates: First submitted 2022-01-18; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Distress; Pain
Keywords: newborn
MeSH Terms: conditions — Dyspnea; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Protocols for the management of end-of-life symptoms — Application of the care protocol and data collection

SUMMARY:
The newborn feels pain and the newborn at the end of life, in the delivery room, is potentially exposed to pain and respiratory distress.

Protocols for the management of end-of-life symptoms in the delivery room are used in current practice with very few validation studies. The protocol used in delivery rooms in Alsace uses fentanyl and midazolam intranasally. It has been used for 3 years and seems to provide satisfactory relief to newborn babies. In doing so, it seems to reassure parents about the quality of support and it seems to meet the expectations of professionals in these anxiety-provoking contexts. Scientific validation of these practices would allow wider dissemination to other maternity teams.

ELIGIBILITY:
Inclusion Criteria:

* Premature or term newborn
* In the delivery room
* In palliative care
* No parental opposition to data collection

Exclusion Criteria:

* Parental refusal or inability to express their consent
* Minor parents
* Very probable survival beyond the delivery room
* Impossibility of giving informed information to the subject (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship or curatorship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature or term newborn in the delivery room
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in pain | 1 day
  Evaluate the effectiveness of the current protocol for the management of pain and discomfort related to end-of-life respiratory distress in newborns receiving palliative care in the delivery room with (Neonatal Facial Coding System) NFCS score
DRFV scores | 1 day
  Presence of DRFV with Silverman score

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KUHN, Principal Investigator — les Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Service de médecine et Réanimation du Nouveau-né - CHU de Strasbourg -France, Strasbourg, Les Hôpitaux Universitaires de Strasbourg
  - Service de pédiatrie - Hôpitaux Civils de Colmar, Colmar
  - Service de pédiatrie - Hôpitaux Civils de Haguenau, Haguenau
  - Service de Néonatologie- Centre Hospitalier de Mulhouse, Mulhouse